CLINICAL TRIAL: NCT01382069
Title: Single Dose, Dose-Ranging and 28-Day Repeat-Dose Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Dimethandrolone Undecanoate (DMAU) in Healthy Men
Brief Title: Phase 1 Study of Dimethandrolone Undecanoate in Healthy Men
Acronym: DMAUPhase1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Washington (Other)
Responsible Party: Principal Investigator, Christina C L Wang, M.D., Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCN010; HHSN275201000080U (Other Grant/Funding Number: NICHD Contract. This is not a grant but a contract)
Record Dates: First submitted 2011-03-25; First posted 2011-06-27 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2016-07

CONDITIONS: Healthy Men; Male Contraception
Keywords: androgen; male contraception; dimethandrolone; healthy men
MeSH Terms: interventions — dimethandrolone-undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Dimethandrolone Undecanoate (Experimental): DMAU group with different doses 100, 200 and 400 groups
  Interventions: Drug: Dimethandrolone Undecanoate

INTERVENTIONS:
Drug: Dimethandrolone Undecanoate — Daily doses of 100, 200 and 400mg of dimethandrolone undecanoate
  Other Names: No other names
  Arms: Dimethandrolone Undecanoate
Drug: Placebo — Placebo with capsules that look like the DMAU capsules but with no active ingredients
  Other Names: no other names
  Arms: Placebo

SUMMARY:
The long term objective is to develop a new male hormone Dimethandrolone Undecanoate (DMAU) as a male hormonal contraceptive.

The study has two parts. The first is a dose escalating study in healthy to assess the safety and tolerability of single dose oral administration of DMAUin healthy men.(Completed)

The second is to study the safety and tolerability of DMAU after 28 days of repeated daily dosing of DMAU in healthy men. (Currently Recruiting) In both parts the investigators will also study the pharmacokinetics of Dimethandrolone (DMA) in the serum after oral administration of DMAU.

DETAILED DESCRIPTION:
The study will be conducted in two centers.

28-Day Repeat-Dose, Dose-Escalation Study: Based on the safety and tolerability of the single dose study and serum DMA levels attained, three doses of two formulations of DMAU were selected for a dose-escalating 28-day repeat dose study. Safety will be assessed in subjects receiving lower dosages before additional men receive higher doses for 28 days. Up to 100 men will be randomized to receive either active drug or an identical number of capsules of placebo. The 24-hour detailed PK of DMA will be assessed on day 1 and 28. Trough levels of DMA will be obtained throughout the 28-day period and at 48 and 72 hours after the last dose. In addition to safety and tolerability, suppression of serum T, gonadotropins, and SHBG will also be assessed as secondary pharmacodynamic (PD) endpoints. Psychosexual diaries for 7 consecutive days and PHQ-9 (questionnaire)will be obtained before and at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening.
2. 18 to 50 years of age.
3. BMI < 33 calculated as weight in kg/ (height in m2 )
4. No history of hormonal therapy use in the last three months prior to the first screening visit.
5. Subject will agree to use a recognized effective method of contraception with his partner (i.e. at a minimum, use double-barrier contraception) during the course of the study treatment and recovery phase.
6. Subjects will refrain from donating blood or plasma during the study period.
7. Subjects will be advised to refrain/abstain from alcoholic beverages and grapefruit juice during the study period.
8. Subjects will not use cannabis or any recreational drugs at least 4 weeks before screening and during the study.
9. In the opinion of the investigator, subject is able to comply with the protocol, understand and sign an informed consent and HIPAA form.
10. Does not meet any of the exclusion criteria.

Exclusion Criteria:

1. Men participating in another clinical trial involving an investigational drug within the last 30 days prior to the first screening visit.
2. Men not living in the catchment's area of the clinic or within a reasonable distance from the study site.
3. Clinically significant abnormal physical and laboratory findings at screening.
4. Elevated PSA (levels ≥ 2.5 ng/mL), according to local laboratory normal values.
5. Abnormal serum chemistry values, according to local laboratory reference ranges that indicate liver or kidney dysfunction or that may be considered clinically significant except for: an upper limit for fasting bilirubin is less than 2 mg/dL, upper limit for cholesterol is less than 220 mg/dL, or upper limit for fasting triglycerides is less than 200 mg/dL.
6. Abnormal semen analyses or abnormal semen concentration as defined by the WHO semen manual.
7. Use of androgens or other body building substances including nutritional supplements within 3 months before first screening visit.
8. Systolic BP > 130 mm Hg and Diastolic blood pressure BP > 80 and mm Hg; ((BP) Blood pressure will be taken 3 times at 5-minute intervals and the mean of all measurements be considered).
9. Clinically significant abnormal EKG and a QTc interval of > 450 msec.
10. PHQ-9 score of 15 or above [for the 28 days study].
11. History of hypertension, including hypertension controlled with treatment.
12. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis.
13. Benign or malignant liver tumors; active liver disease.
14. History of breast carcinoma.
15. Known history of androgen deficiency due to hypothalamic-pituitary or testicular disease.
16. Known history of cardiac, renal, hepatic or prostatic disease.
17. Positive serology for Hepatitis or HIV at screening visit.
18. A serious systemic disease such as diabetes mellitus or obesity (body weight greater than BMI >33 kg/m2 as above).
19. History of known, untreated sleep apnea.
20. Known or suspected alcoholism or drug abuse that may affect metabolism/transformation of steroid hormones and study treatment compliance.
21. Partner is known to be pregnant.
22. Men desiring fertility within the first 24 weeks of study participation.
23. Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine will be advised of the relative and temporary hazards that participating in this study may have for their fertility or sporting status.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Single Dose, Dose-Ranging and 28-Day Repeat-Dose Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Dimethandrolone Undecanoate (DMAU) in Healthy Men | 1 day
  Number of severe or serious adverse event fdter escalating single doses of Dimethandrolone Undecanoated in a single dose escalating study or after 28 days repeat dosing in healthy men

SECONDARY OUTCOMES:
Single Dose, Dose-Ranging and 28 days Repeat Dose Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Dimethandrolone Undecanoate (DMAU) in Healthy Men | 28 days
  Serum Dimethandrolone Levels on day 28
Single Dose, Dose-Ranging and 28-Day Repeat-Dose Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Dimethandrolone Undecanoate (DMAU) in Healthy Men | 2 days Food or no food
  Serum Dimethandrolone levels
Single Dose, Dose-Ranging and 28-Day Repeat-Dose Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics Study of Dimethandrolone Undecanoate (DMAU) in Healthy Men | 28 DAYS
  Serum hormone levels (Testosterone (T), FSH and LH and SHBG) and sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center; Stephanie Page, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute, Torrance, California
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Attardi BJ, Hild SA, Reel JR. Dimethandrolone undecanoate: a new potent orally active androgen with progestational activity. Endocrinology. 2006 Jun;147(6):3016-26. doi: 10.1210/en.2005-1524. Epub 2006 Feb 23. PMID 16497801
- [Background] Attardi BJ, Engbring JA, Gropp D, Hild SA. Development of dimethandrolone 17beta-undecanoate (DMAU) as an oral male hormonal contraceptive: induction of infertility and recovery of fertility in adult male rabbits. J Androl. 2011 Sep-Oct;32(5):530-40. doi: 10.2164/jandrol.110.011817. Epub 2010 Dec 16. PMID 21164142
- [Background] Attardi BJ, Marck BT, Matsumoto AM, Koduri S, Hild SA. Long-term effects of dimethandrolone 17beta-undecanoate and 11beta-methyl-19-nortestosterone 17beta-dodecylcarbonate on body composition, bone mineral density, serum gonadotropins, and androgenic/anabolic activity in castrated male rats. J Androl. 2011 Mar-Apr;32(2):183-92. doi: 10.2164/jandrol.110.010371. Epub 2010 Aug 26. PMID 20798389
- [Derived] Yuen F, Thirumalai A, Fernando FA, Swerdloff RS, Liu PY, Pak Y, Hull L, Bross R, Blithe DL, Long JE, Page ST, Wang C. Comparison of metabolic effects of the progestational androgens dimethandrolone undecanoate and 11beta-MNTDC in healthy men. Andrology. 2021 Sep;9(5):1526-1539. doi: 10.1111/andr.13025. Epub 2021 May 22. PMID 33908182
- [Derived] Thirumalai A, Yuen F, Amory JK, Hoofnagle AN, Swerdloff RS, Liu PY, Long JE, Blithe DL, Wang C, Page ST. Dimethandrolone Undecanoate, a Novel, Nonaromatizable Androgen, Increases P1NP in Healthy Men Over 28 Days. J Clin Endocrinol Metab. 2021 Jan 1;106(1):e171-e181. doi: 10.1210/clinem/dgaa761. PMID 33090208
- [Derived] Thirumalai A, Ceponis J, Amory JK, Swerdloff R, Surampudi V, Liu PY, Bremner WJ, Harvey E, Blithe DL, Lee MS, Hull L, Wang C, Page ST. Effects of 28 Days of Oral Dimethandrolone Undecanoate in Healthy Men: A Prototype Male Pill. J Clin Endocrinol Metab. 2019 Feb 1;104(2):423-432. doi: 10.1210/jc.2018-01452. PMID 30252061
- [Derived] Ayoub R, Page ST, Swerdloff RS, Liu PY, Amory JK, Leung A, Hull L, Blithe D, Christy A, Chao JH, Bremner WJ, Wang C. Comparison of the single dose pharmacokinetics, pharmacodynamics, and safety of two novel oral formulations of dimethandrolone undecanoate (DMAU): a potential oral, male contraceptive. Andrology. 2017 Mar;5(2):278-285. doi: 10.1111/andr.12303. Epub 2016 Dec 1. PMID 27907978